CLINICAL TRIAL: NCT01912131
Title: Person-Centered Oncology Care and Choices (P-COCC): Piloting and Initial Randomized Testing of a Combined Values Narrative Interview and Video Education Advance Care Planning Program in Gastrointestinal Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-120
Record Dates: First submitted 2013-07-25; First posted 2013-07-30 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastrointestinal Cancer
Keywords: 13-120
MeSH Terms: interventions — Patient Care Planning; Videotape Recording

ARMS (4):
- First 24 patients Cognitive interviewing (Experimental): Part 1 - This first study phase will involve interviewing 24 patients to ask for their feedback on the appropriateness of questions being developed for use in the narrative interviewing in part 2 of the study. The cognitive interview will be audio-recorded. Demographics and ECOG performance status will be recorded prior to the cognitive interview.
  Interventions: Behavioral: single pilot interview
- usual care (Active Comparator): As outlined ECOG performance status will be recorded at the time of registration without the subject's involvement. Quality of life, treatment satisfaction, distress and peacefulness will also be recorded at baseline. Subjects will neither be shown the goals-of-care (GOC) video nor undergo the narrative interview process - they will be contacted as per re-assessment.
  Interventions: Behavioral: usual care; Behavioral: Part 2
- video-only arm (Experimental): As outlined ECOG performance status will be recorded at the time of registration without the subject's involvement. Quality of life, treatment satisfaction, distress and peacefulness will also be recorded at baseline. Subjects will be shown the goals-of-care (GOC) video but not undergo a narrative interview process - they will be contacted as per re-assessment.
  Interventions: Behavioral: goals-of-care (GOC) video; Behavioral: Part 2
- combined narrative and video (P-COCC) arm (Experimental): As outlined ECOG performance status will be recorded at the time of registration without the subject's involvement. Quality of life, treatment satisfaction, distress and peacefulness will also be recorded at baseline. subjects will watch the goals-of-care (GOC) video (described in detail in the next paragraph) and then be given the narrative question stem vetted/assessed in part 1 including any changes made to that stem in the process of Part 1 testing. Subjects in P-COCC arm will then be contacted for a telephone interview and audio-taping of their narrative. Interviews will be semi- structured and based off the narrative stem that subjects were previously given for review. Interviews will last approximately 30-45 minutes and will be conducted by staff from the MSKCC Department of Psychiatry & Behavioral Sciences.
  Interventions: Behavioral: goals-of-care (GOC) video and narrative question; Behavioral: Part 2

INTERVENTIONS:
Behavioral: single pilot interview — Part 1 participants will be scheduled for their single pilot interview. There are no additional assessments.
  Arms: First 24 patients Cognitive interviewing
Behavioral: goals-of-care (GOC) video — Subjects will be shown the goals-of-care (GOC) video but not undergo a narrative interview process - they will be contacted as per re-assessment.
  Arms: video-only arm
Behavioral: goals-of-care (GOC) video and narrative question — subjects will watch the goals-of-care (GOC) video (described in detail in the next paragraph) and then be given the narrative question stem vetted/assessed in part 1 including any changes made to that stem in the process of Part 1 testing. Subjects in P-COCC arm will then be contacted for a telephone interview and audio-taping of their narrative. Interviews will be semi- structured and based off the narrative stem that subjects were previously given for review. Interviews will last approximately 30-45 minutes and will be conducted by staff from the MSKCC Department of Psychiatry & Behavioral Sciences,
  Arms: combined narrative and video (P-COCC) arm
Behavioral: usual care — Subjects in the usual care arm will neither be given the narrative stem nor watch the video.
  Arms: usual care
Behavioral: Part 2 — Will be a proof-of-concept, small scale, RCT to measure P-COCC acceptability and other quantitative and qualitative effects. Seventy five participants will be randomized to Usual Care, Video, or Video and Interview.
  Arms: combined narrative and video (P-COCC) arm; usual care; video-only arm

SUMMARY:
This study is being done to get individuals' feedback on advanced care planning and decision making.

This study is divided into two parts (Part 1 and Part 2). The purpose of Part 1 is to survey people to find out what is important to people with advanced cancer (again, their values, such as their goals, concerns and sources of support). This has never been done before in the way the investigators are doing it, and that is why this is called a "pilot" study, which is where a new method or treatment is being created and evaluated.

The purpose of Part 2 is to see if combining a medical options video with a short interview about values helps people with how they feel about their medical situation, and what they know about their medical options for their medical situation.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read and understand English well enough to complete study assessments and interviews in the judgement of the consenting professional
* 18 years of age and older
* Be seen regularly (at least monthly) at an MSKCC GI medical oncology clinic
* Has an exocrine GI cancer with MSKCC pathology confirmation at the primary or metastatic anatomic site
* Non-metastatic GI cancers are eligible only if the Eastern Cooperative Oncology Group (ECOG) performance status54 is 2,3, or 4 at the time of consent (although patients with locally advanced [stage III] and inoperable pancreatic cancers are eligible regardless of their performance status)
* Has a metastatic neuroendocrine histology with MSKCC pathology confirmation as moderately or poorly differentiated or intermediate or high grade
* A referring physician's estimate of patient life expectancy must be between 1-12 months. We use this life expectancy range in order to ensure some degree of subject homogeneity for the purpose of sample size and methodologic design. Also, these timeframes were chosen in order to test an intervention in patients with serious illness (under 1 year prognosis).
* Part 2 Only: Did not complete Part 1 of the study.

Exclusion Criteria:

* Short Portable Mental Status Questionnaire (SPMSQ) score of less than "intact mental functioning" (3 or more errors).
* Significant psychiatric or cognitive disturbance sufficient, in the consenting professional's or investigator's judgment, to preclude providing informed consent or participating in the interventions (i.e., acute psychiatric symptoms which require individual treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
assess the acceptability of this piloted P-COCC intervention | 2 years
  primary outcome is assessed in Part 2 of the study, and is acceptability of this newly- developed P-COCC intervention, as measured by subjects in P-COCC arm who will complete three Likert scale questions examining the degree to which they found the narrative recording process.

SECONDARY OUTCOMES:
quantitative analyses | 2 years
  pre-post scoring on our various psychometric questionnaires (quantitative) and of the subject responses during narrative interviewing (qualitative)
qualitative analyses | 2 years
  pre-post scoring on our various psychometric questionnaires (quantitative) and of the subject responses during narrative interviewing (qualitative)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Epstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/